CLINICAL TRIAL: NCT05205226
Title: Efficacy and Safety of Local Radiotherapy for Residual Tumor Lesions During the First-line Treatment of Advanced Non-small Cell Lung Cancer: a Retrospective-real World Study
Brief Title: Local Radiotherapy for Residual Tumor Lesions During the First-line Treatment
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Other Study IDs: SPLENDOR
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2018-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to confirmed that local radiotherapy for residual lesions can significantly prolong the efficacy of chemotherapy combined with immunotherapy in the initial treatment of advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥18，Advanced Non-small Cell Lung Cancer Confirmed by Histopathology Patients received platinum-based chemotherapy combined with immunotherapy

Exclusion Criteria:

* EGFR/ALK/ROS1 driver gene mutation
* Chemotherapy only
* Concurrent radio-chemotherapy
* Surgery
* Single-agent immunotherapy
* No treatment information available

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with non driver mutation advanced non-small-cell lung cancer non driver mutation
Sampling Method: Probability Sample
Enrollment: 636 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
PFS | January 2018 to June 2021
  Progression free survival time

SECONDARY OUTCOMES:
RT | January 2018 to June 2021
  radiotherapy control time

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang C Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China